CLINICAL TRIAL: NCT06935552
Title: Ketamine and Lidocaine Infusion for Refractory Chronic Migraine: Comparative Study
Brief Title: Ketamine and Lidocaine Infusion in Refractory Chronic Migraine
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AbdElRahman Mohamed Mohamed Mohamed, Resident doctor in neurology and psychiatry department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ketamine vs lidocaine in RCM
Record Dates: First submitted 2025-04-07; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Refractory Chronic Migraine
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine (Experimental): will receive ketamine
  Interventions: Drug: Ketamine infusion
- Lidocaine (Experimental): will receive lidocaine
  Interventions: Drug: Lidocaine Intravenous Infusion
- Dextrose (Placebo Comparator)
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Ketamine infusion — group A will receive ketamine intravenous infusion
  Arms: Ketamine
Drug: Lidocaine Intravenous Infusion — group B will receive lidocaine intravenous infusion
  Arms: Lidocaine
Drug: Dextrose 5% in water — group C will only receive Dextrose 5% in water
  Arms: Dextrose

SUMMARY:
Ketamine and lidocaine infusion for refractory chronic migraine: Comparative Study

ELIGIBILITY:
Inclusion Criteria:

* All participants must fulfill the following inclusion criteria

  1. medically stable outpatients with confirmed diagnosis of refractory chronic migraine according to American Headache society
  2. Are reliable and willing to make themselves available for the duration of the study and are willing to follow up.
  3. Men or women older than 18years of age.
  4. clear written informed consent from each participant in the trial.
  5. Adult patients with refractory migraine or refractory chronic migraine defined according to the American headache society

Exclusion Criteria:

1. Pregnancy, active psychosis, liver disease, uncontrolled cardiac disease or cardiac rhythm abnormalities
2. presence of clinically significant medical or psychiatric condition that may increase the risk associated with the study
3. participation in any other type of medical research that may interfere with the interpretation of the study.
4. patients with hemocoagulation disorders, local infection or those who refused to consent

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pain scale using Numeric rating scale | From enrollment to the end of treatment at 6 weeks
  Pain assessment by using a Numeric rating scale (0 (no pain) to 10 (worst possible pain). Scores of 1-3 are considered mild, 4-6 moderate, and 7-10 severe) before the infusion and daily for 1-week post infusion, then weekly for 6 weeks post infusion
Changes in pain scale using Migraine disability assessment | From enrollment to the end of treatment at 6 weeks
  Migraine disability assessment test before the infusion and daily for 1-week post infusion, then weekly for 6 weeks post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nageh Fouly Kamel, PhD., Study Chair — Assiut University; Mohamed Ahmed Abdelhameed, PhD., Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schulman EA, Lake AE 3rd, Goadsby PJ, Peterlin BL, Siegel SE, Markley HG, Lipton RB. Defining refractory migraine and refractory chronic migraine: proposed criteria from the Refractory Headache Special Interest Section of the American Headache Society. Headache. 2008 Jun;48(6):778-82. doi: 10.1111/j.1526-4610.2008.01132.x. Epub 2008 May 14. PMID 18484982
- [Background] Ray JC, Cheng S, Tsan K, Hussain H, Stark RJ, Matharu MS, Hutton E. Intravenous Lidocaine and Ketamine Infusions for Headache Disorders: A Retrospective Cohort Study. Front Neurol. 2022 Mar 9;13:842082. doi: 10.3389/fneur.2022.842082. eCollection 2022. PMID 35356451
- [Background] Lauretti GR. Mechanisms of analgesia of intravenous lidocaine. Rev Bras Anestesiol. 2008 May-Jun;58(3):280-6. doi: 10.1590/s0034-70942008000300011. English, Portuguese. PMID 19378524
- [Background] Kohrs R, Durieux ME. Ketamine: teaching an old drug new tricks. Anesth Analg. 1998 Nov;87(5):1186-93. doi: 10.1097/00000539-199811000-00039. No abstract available. PMID 9806706
- [Background] Natoli JL, Manack A, Dean B, Butler Q, Turkel CC, Stovner L, Lipton RB. Global prevalence of chronic migraine: a systematic review. Cephalalgia. 2010 May;30(5):599-609. doi: 10.1111/j.1468-2982.2009.01941.x. PMID 19614702